CLINICAL TRIAL: NCT01106469
Title: Single and Multiple Ascending Dose Study to Investigate the Safety, Tolerability, Food Effect, Pharmacokinetics, and Pharmacodynamics of JNJ-41443532 in Healthy Male Subjects
Brief Title: Pharmacokinetics (PK) and Pharmacodynamics (PD) Study of Single and Multiple Ascending Doses of JNJ-41443532 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: CR017065; 41443532EDI1001 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.)
Record Dates: First submitted 2010-04-15; First posted 2010-04-20 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Healthy
Keywords: Healthy Volunteers; Healthy; JNJ-41443532; Pharmacokinetics
MeSH Terms: interventions — JNJ-41443532

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (7):
- 001 (Experimental): JNJ-41443532 25mg tablet once daily
  Interventions: Drug: JNJ-41443532
- 002 (Experimental): JNJ-41443532 100mg tablet once daily
  Interventions: Drug: JNJ-41443532
- 003 (Experimental): JNJ-41443532 250mg tablet once daily
  Interventions: Drug: JNJ-41443532
- 004 (Experimental): JNJ-41443532 500mg once daily (with 250mg tablets)
  Interventions: Drug: JNJ-41443532
- 005 (Experimental): JNJ-41443532 1000mg once daily (with 250mg tablets)
  Interventions: Drug: JNJ-41443532
- 006 (Experimental): JNJ-41443532 1500mg once daily (with 250mg tablets)
  Interventions: Drug: JNJ-41443532
- 007 (Placebo Comparator): Placebo Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-41443532 — 25mg tablet once daily
  Arms: 001
Drug: JNJ-41443532 — 250mg tablet once daily
  Arms: 003
Drug: JNJ-41443532 — 1500mg once daily (with 250mg tablets)
  Arms: 006
Drug: JNJ-41443532 — 100mg tablet once daily
  Arms: 002
Drug: JNJ-41443532 — 1000mg once daily (with 250mg tablets)
  Arms: 005
Drug: Placebo — Matching placebo
  Arms: 007
Drug: JNJ-41443532 — 500mg once daily (with 250mg tablets)
  Arms: 004

SUMMARY:
The purpose of this study is to investigate the safety, tolerability, food effect as well as the pharmacokinetics (how the drug is absorbed in the body, how it is distributed within the body and how it is removed from the body over time) and pharmacodynamics (the effects of the drug) of single and multiple ascending doses of JNJ-41443532 in healthy male participants.

DETAILED DESCRIPTION:
This is a randomized (study drug assigned by chance), double-blind (neither physician nor participant knows the name of the assigned drug), placebo-controlled, single and multiple ascending dose study conducted at a single study center. The study has 4 parts. Part 1 is a randomized, double-blind, alternating panel, single ascending oral dose study. Two alternating treatment panels (A and B) each with nine healthy male participants will be studied with successively increasing dose levels. Part 2 is a randomized, open-label (all people involved know the identity of the intervention), 2-period crossover study to evaluate what the effect of administering JNJ- 41443532 with food (i.e. standard high fat breakfast meal) relative to administration in the fasted state will have on pharmacokinetics/blood levels of JNJ-41443532. Part 3 is a randomized, double-blind, single oral dose study in obese, otherwise healthy male participants. Part 4 is a double-blind, randomized, placebo-controlled multiple ascending dose study in up to 5 sequential treatment groups of healthy male participants. Safety assessments include monitoring of adverse events, and evaluation of lab results, cardiac parameters, vital signs, and physical exams. In Parts 1, 2, and 3 participants receive study medication (JNJ-41443532 or placebo) orally on Day 1 after an overnight fast of at least 10 hours; planned doses are 25 to 1500 mg. In Part 4, participants receive study medication (JNJ-41443532 or placebo) orally each day for 10 consecutive days after an overnight fast of at least 10 hours; planned doses are 100 to 1000 mg.

ELIGIBILITY:
Inclusion Criteria:

* Males, age 18 to 45 years inclusive for Part 1 and age 18 to 55 years inclusive for Parts 2, 3, and 4
* Weight = 60 kilograms and Body Mass Index (BMI) between 18.5 and 29.9 kg/m2 (inclusive)
* BMI between 30 to 39.9 kg/m2 for obese participants
* Healthy on the basis of physical examination, medical history, vital signs, electrocardiogram (ECG), and clinical laboratory tests performed at screening
* Men must agree to use a double barrier method of birth control (e.g. condom and use of spermicide with diaphragm, hormonal contraceptives or intrauterine devices by female partner) and to not donate sperm during the study and for 3 months after receiving the last dose of study drug
* Willing to adhere to the prohibitions and restrictions specified in this protocol

Exclusion Criteria:

* History of, or currently active, significant illness or medical disorders, including (but not limited to) cardiovascular disease (including cardiac arrhythmias, myocardial infarction, stroke, peripheral vascular disease), endocrine or metabolic disease (e.g. hyper/hypo-thyroidism), hematological disease (e.g. von Willebrand's disease or other bleeding disorders), respiratory disease, hepatic or gastrointestinal disease, neurological or psychiatric disease, ophthalmologic disorders (including retinal disorders or cataracts), neoplastic disease, skin disorder, or any other illness that the Investigator considers should exclude the participant
* Participants at risk for QTc prolongation (specific heart rhythm irregularity)
* Within 12 months prior to screening, has had a clinically important, serious infection (e.g. hepatitis, pneumonia, or pyelonephritis), has been hospitalized for an infection or has been treated with intravenous (IV) antibiotics for an infection
* Smoker or tobacco user within the past 3 months
* History of alcohol or drug abuse
* History of clinically significant drug and/or food allergies, including allergies or intolerance (e.g. lactose intolerance)
* Donation of 1 or more units of blood or acute loss of an equivalent amount of blood within 60 days prior to study drug administration
* Received an experimental drug or used an experimental medical device within 60 days

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2010-02; Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Determine the pharmacokinetic properties of single and multiple doses JNJ-41443532 as determined by blood level concentrations. | Part 1 - Approximately 13 weeks; Part 2 - Approximately 7 weeks; Part 3 - Approximately 6 weeks; Part 4 - Approximately 7 weeks

SECONDARY OUTCOMES:
Determine the safety and tolerability of JNJ-41443532 as determined by evaluation of adverse events, lab results, cardiac monitoring, vital signs, and physical exams. | Part 1 - Approximately 13 weeks; Part 2 - Approximately 7 weeks; Part 3 - Approximately 6 weeks; Part 4 - Approximately 7 weeks
To explore the relationship between JNJ-41443532 plasma concentrations and pharmacodynamic effects (concentration-effect relationships). | Part 1 - Approximately 13 weeks; Part 2 - Approximately 7 weeks; Part 3 - Approximately 6 weeks; Part 4 - Approximately 7 weeks
To explore the pharmacodynamic (PD) effects of JNJ-41443532 and to compare the differences between treatment groups | Part 1 - Approximately 13 weeks; Part 2 - Approximately 7 weeks; Part 3 - Approximately 6 weeks; Part 4 - Approximately 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- Merksem, Belgium